CLINICAL TRIAL: NCT00159016
Title: The Possible Role of Glivec in Patients With Tumor Cells Positive for C-kit or Platelet Derived Growth Factor Receptor (PDGFR); a Multi Center Study.
Brief Title: Role of Glivec in Patients With Tumor Cells Positive for C-kit or PDGFR; a Multi Center Study.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: the PI is no longer work at Hadassah
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 291004-HMO-CTIL
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2011-04-28 (Estimated); Status verified 2005-09

CONDITIONS: Metastatic Solid Tumors.
MeSH Terms: interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: Glivec

SUMMARY:
This is a phase II, multi-center (Israeli), open label, non-randomized trial for every patient with the specified tumors expressing c-kit or PDGFR. Expression of these kinases will be investigated in tumor samples obtained at the time of diagnosis or from the time of recurrent disease. Every patient with positive expression of either of the kinases will be evaluated for quantitative and qualitative evidence of disease prior to entry into the study, and if possible, no other treatment will be given concomitantly, to allow evaluation of the net effect of Glivec on tumor growth kinetics, searching for measurable evidence of response.

Glivec is supplied to the study investigators by Novartis Pharmaceutical. Patients will receive Glivec 400mg-800mg p.o./day for an exposure period of up to 12 months provided that in the opinion of the investigator the patient is benefiting from treatment with Glivec, and in the absence of any safety concern. For patients with brain tumors who are not receiving concomitant enzyme inducing anti-convulsant drugs, the recommended dose of Glivec is 800mg/day.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age.
* Histologically documented diagnosis of one of the specified tumors, which is malignant as well as unresectable and/or metastatic and therefore, incurable with any conventional multimodality approach and immunohistochemical documentation of c-kit (CD117) or PDGFR expression in the primary tumor or metastases by tumor (preferably on a tumor sample taken within 6 week of study entry).
* At least one measurable site of disease as defined by Southwestern Oncology Group Solid Tumor Response Criteria.
* Female patients of child-bearing potential must have negative pregnancy test.
* Signed informed consent form.
* Life expectancy >3 months.

Exclusion Criteria:

* Patient has received any other investigational agents within 28 days of the first day of study drug dosing.
* Existence of any evidence of another malignant disease, except superficial non-melanoma skin cancer.
* Patient has a known brain metastases.
* Patient previously received radiotherapy to >25% of the bone marrow.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2002-08; Study Completion 2005-09

PRIMARY OUTCOMES:
Evaluate activity of Glivec in escalating doses 400 up to 800mg/day in patients with a large variety of metastatic solid tumors expressing c-kit or PDGFR.

SECONDARY OUTCOMES:
Evaluate the toxicity of Glivec in patients with solid tumors.

CONTACTS AND LOCATIONS:
Overall Officials: Shimon Slavin, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel